CLINICAL TRIAL: NCT06576180
Title: Effects of Neoadjuvant Therapy With Carboplatin, Paclitaxel Combined With Anti-PD-1 Drugs on Cognitive Function in Patients With Resectable Head and Neck Squamous Cell Carcinoma: a Prospective Cohort Study
Brief Title: Effects of Neoadjuvant Therapy With Carboplatin, Paclitaxel Combined With Anti-PD-1 Drugs on Cognitive Function in Patients With Resectable Head and Neck Squamous Cell Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Song Fan, MD, Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSKY-2024-647-01
Record Dates: First submitted 2024-08-23; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Neoadjuvant therapy+ Surgery group( Group A): The patient was diagnosed with head and neck squamous cell carcinoma (stage I-IVA), untreated, and planned to undergo surgical treatment + combined chemotherapy and immunotherapy.
  Interventions: Drug: Carboplatin（ neoadjuvant）; Drug: Paclitaxel （neoadjuvant）; Drug: Anti-PD-1 Drugs; Procedure: Surgical resection
- Direct surgery group (Group B): The patient was diagnosed with head and neck squamous cell carcinoma (stage I-IVA), untreated, and planned to undergo surgery.
  Interventions: Procedure: Surgical resection
- Healthy people (Group C): Healthy people

INTERVENTIONS:
Drug: Carboplatin（ neoadjuvant） — Carboplatin (IV), AUC=5，administered by intravenous (IV) infusion on Day 1 of each 21-day cycle
  Groups: Neoadjuvant therapy+ Surgery group( Group A)
Drug: Paclitaxel （neoadjuvant） — Paclitaxel 260mg/m2 administered by intravenous (IV) infusion on Day 1 of each 21-day cycle
  Groups: Neoadjuvant therapy+ Surgery group( Group A)
Drug: Anti-PD-1 Drugs — Anti-PD-1 Drugs 200 mg administered by intravenous (IV) infusion on Day 1 of each 21-day cycle
  Groups: Neoadjuvant therapy+ Surgery group( Group A)
Procedure: Surgical resection — Standard of care
  Groups: Direct surgery group (Group B); Neoadjuvant therapy+ Surgery group( Group A)

SUMMARY:
The goal of this observational study is to learn about the Effects of neoadjuvant therapy with carboplatin, paclitaxel combined with anti-PD-1 drugs on cognitive function in patients with resectable head and neck squamous cell carcinoma: a prospective cohort study

ELIGIBILITY:
Inclusion Criteria:

* 1: The patient was diagnosed with head and neck squamous cell carcinoma (stage I-IVA), without treatment, and planned to undergo only surgical treatment or surgical treatment + chemotherapy and immunotherapy.

  2: Can speak Chinese and have certain reading and writing skills

  3: Healthy group: Dental inpatients with non-oral cancer, no history of neurological diseases, and no previous history of malignant tumors

Exclusion Criteria:

* 1: Brain tumor, brain injury, or stroke at baseline or during follow-up

  2: A history of stroke or a medical condition that puts you at high risk for future dementia or recurrence

  3: Active mental illness or active narcotic drug use, including using alcohol more than 4 times per day or more than 4 times per week

  4: Neurocognitive diseases that affect cognitive function, such as Parkinson's disease or Alzheimer's disease

  5: History of drug-associated encephalopathy or brain infection

  6: Patients who change their treatment plan during treatment

  7: Patients who are currently taking or have taken antidepressants

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patients were diagnosed with head and neck squamous cell carcinoma (stages I-IV) and did not receive treatment. They planned to receive only surgical treatment or combined surgical treatment + chemotherapy and immunotherapy. They were divided into two groups, and the participating groups were selected according to the inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 306 (Estimated)
Dates: Start 2024-08-23 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
cognitive adverse events, CoAE | Baseline, 9 weeks, 6 months, 12 months
  Scores on two or more of the neuropsychological battery tests (NBT) of the HVLT-R, COWA, and TMT are 1.5 SD below the standard mean (or the mean score of an appropriate control group), Or a single test score that is 2.0 SD below the mean can be marked as an objective cognitive adverse event (CoAE).

SECONDARY OUTCOMES:
Major pathological response rate | Within 30 days after surgery
  Defined as the proportion of subjects with ≤10% viable tumor cells in resection specimens to total subjects
Montreal Cognitive Assessment, MoCA | The total score is obtained by adding up the scores of each item, and the full score is 30 points. The application results of the original English version of the scale designer show that if the number of years of education is ≤12 years, 1 point is added,
  Baseline, 9 weeks, 6 months, 12 months
perceived cognitive decline events , PCDE | 1/2 standard deviation (SD) of the PCI score in the baseline healthy population is defined as a minimal clinically important difference (MCID), and a change in PCI score that exceeds the MCID in each test will be labeled as PCDE.
  Baseline, 9 weeks, 6 months, 12 months
complete pathological response rate | Within 30 days after surgery
  Defined as the proportion of subjects without viable tumor cells in the resection specimen to the total subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guanzhou, Guangdong, China